CLINICAL TRIAL: NCT00934128
Title: An Exploratory Trial of Bilevel Positive Airway Pressure Device and High Flow Oxygen for Persistent Dyspnea in Advanced Cancer Patients
Brief Title: High Flow Oxygen and Bilevel Airway Pressure for Persistent Dyspnea in Patients With Advanced Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0164
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancer; Persistent Dyspnea; Shortness of breath; Specialized breathing devices; Bilevel positive airway pressure device; BIPAP; High flow oxygen delivery device; VapoTherm; Edmonton Symptom Assessment Scale; ESAS
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: BiPAP then Vapotherm (Experimental): Bilevel positive airway pressure device (BiPAP) then Vapotherm air delivery.
  Interventions: Device: Vapotherm; Device: BIPAP
- Group 2: Vapotherm then BiPAP (Experimental): Vapotherm air delivery then BiPAP.
  Interventions: Device: Vapotherm; Device: BIPAP

INTERVENTIONS:
Device: Vapotherm — Deliver air in and out of the lungs, warmed, filtered for bacteria, and then delivered through the nose using a tube under the nostrils.
  Other Names: High flow oxygen delivery system
Device: BIPAP — Air given through a mask, and amount can be set to different levels allowing more air in and out of lungs without using as much effort as regular breathing.
  Other Names: Bilevel positive airway pressure device

SUMMARY:
The goal of this clinical research study is to learn if specialized breathing devices reduce the sensation of shortness of breath in patients with advanced cancer who are experiencing shortness of breath. Researchers want to learn if these devices can help to control shortness of breath.

The 2 devices being tested and compared are called BiPAP (bilevel positive airway pressure) and Vapotherm.

DETAILED DESCRIPTION:
Study Devices:

The BiPAP device is designed to help people get more air in and out of their lungs without using as much effort as regular breathing. The air is given through a mask, and the amount of air can be set to different levels.

The Vapotherm device is also designed to deliver air in and out of the lungs. The air is warmed, filtered for bacteria, and then delivered through the nose using a tube under the nostrils.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups.

* Group 1 will receive air through BiPAP for up to 2 hours and then air through Vapotherm for up to 2 hours.
* Group 2 will receive air through Vapotherm for up to 2 hours and then air through BiPAP for up to 2 hours.

The study staff will help you use the devices.

If you have trouble with one of the devices, you can be switched to the other device before the 2-hour period is over.

After using the first device, you will wait for up to 60 minutes before switching over to the other device. This waiting period will occur no matter if you used the first device for the full 2 hours or not.

During the waiting period, you will return to the same air delivery device and oxygen level that you were using just before you started the study. The study staff will also be checking to see if you are still eligible to use the second device.

Study Tests:

During the study period, your vital signs and level of air breathed out will be recorded using a measuring device on your chest.

Before and after using the devices, you will rate how hard it is to catch your breath.

After using the second device, you will fill out a questionnaire that has questions about which device you prefer. This should take less than 5 minutes.

Length of Study:

You will be on this study for up to 5 hours. You will be taken off study and the device will be stopped if intolerable side effects occur while using a study device.

Use of Other Drugs:

During the 4-5 hour study period, you will not be allowed to take certain drugs for standard care that may affect the study tests. These drugs include certain pain-killer drugs (such as morphine and hydromorphone), steroids (such as prednisone and dexamethasone), and inhaled drugs (such as ipratropium and salbutamol).

Any doses of inhaled drugs (regularly scheduled doses and "as needed" doses) and any "as needed" doses of pain-killer drugs and steroids that fall within the 4-5 hour study period will be put on hold and will be given to you right after the study is complete.

You may, however, choose to take these drugs, either because your shortness of breath is not controlled, or because these drugs are needed to treat other problems (such as pain). If you and your doctor decide that you should take these drugs during the study period, you will be taken off study so you can receive these drugs. The reason for stopping your study participation is that these drugs may affect how you rate your shortness of breath.

This is an investigational study. The BIPAP and Vapotherm devices are commercially available and FDA approved for delivering oxygen when medically needed, including in patients with advanced cancer. The investigational part of this study is to collect information from asking patients to rate how well the study devices may affect shortness of breath.

Up to 50 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. History of advanced cancer, defined as locally advanced, recurrent or metastatic disease
2. Patients with persistent dyspnea, defined in this study as dyspnea at rest with an average intensity level >/=3 out of a Numeric Rating Scale from 0 to 10 for at least 2 week and just prior to study initiation, despite supplemental oxygen of up to 21 L/min to keep oxygen saturation >/=90%
3. Dyspnea is judged clinical to be predominantly due to underlying malignancy, with or without obstructive lung disease
4. Inpatient at MD Anderson Cancer Center
5. Patients with cancer treatment related dyspnea are eligible for this study if they meet the eligibility criteria above.
6. Able to communicate in English
7. Expected life expectancy >1 week
8. Patients with a diagnosis of pneumonia are also eligible for this study if they meet the eligibility criteria above, with dyspnea >=2 weeks prior to the diagnosis of pneumonia.
9. Age 18 or greater

Exclusion Criteria:

1. Patients who remain hypoxic (i.e. O2 saturation <90% despite maximal oxygen delivery (21 L/min) are not included in this study because they are considered to have severe life-threatening respiratory failure and are too unstable for study inclusion.
2. Hemodynamic instability (Heart Rate (HR) >140, systolic blood pressure (SBP) <80) within 24 hours of study initiation (as per Clinic Station)
3. Acute respiratory distress requiring intubation
4. Delirium as indicated by a Memorial Delirium Assessment Scale (MDAS) of 13 or higher
5. Glasglow coma scale <8
6. Excessive airway secretions interfering with BIPAP administration
7. History of facial trauma within 1 month of enrollment
8. Upper GI bleed within 2 weeks of enrollment or esophageal rupture
9. Partial or complete small bowel obstruction or severe nausea/vomiting (ESAS nausea >7/10) within 48 hours of enrollment
10. Hemoglobin <8 g/dL at the time of enrollment (blood draw within last 2 weeks)
11. Acute exacerbation of COPD or CHF within 2 weeks of enrollment by history or physical
12. Unwilling to provide informed consent
13. Diagnosis of non-cancer related dyspnea (e.g. Chronic obstructive pulmonary disease (COPD), congestive heart failure (CHF) or any chronic respiratory disease) requiring supplemental home oxygen prior to hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period August 2009 to February 2012. All recruitment was done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Group 1: BiPAP Then Vapotherm: Bilevel positive airway pressure device (BiPAP) then high flow oxygen (HFO) delivery using Vapotherm device.
Period: First Intervention (2 Hours)
Arm/Group | Group 1: BiPAP Then Vapotherm | Group 2: Vapotherm Then BiPAP
Started | 15 | 15
Completed | 10 | 13
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 4 | 1
Not completed — Treatment Delivery Order Switched | 1 | 0
Period: Washout Period (1 Hour)
Arm/Group | Group 1: BiPAP Then Vapotherm | Group 2: Vapotherm Then BiPAP
Started | 10 | 13
Completed | 3 | 8
Not Completed | 7 | 5
Not completed — Patient preference | 1 | 3
Not completed — Pain | 1 | 0
Not completed — Too tired | 1 | 0
Not completed — Dyspnea too low to continue | 4 | 2
Period: Second Intervention (2 Hours)
Arm/Group | Group 1: BiPAP Then Vapotherm | Group 2: Vapotherm Then BiPAP
Started | 3 | 8
Completed | 3 | 5
Not Completed | 0 | 3
Not completed — Claustrophobia/anxiety | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: BiPAP Then Vapotherm | Group 2: Vapotherm Then BiPAP | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Full Range); unit: years] | 63 [47 to 79] | 59 [29 to 79] | 61 [29 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 9 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing Study Intervention
Description: Retention rate defined as the percentage of subjects able to complete the first phase (washout) of study.
  A variable washout/follow-up period after the first intervention was used to determine the optimal duration required for participants to return to baseline dyspnea level. After participants completed the first intervention by one hour, they were able to proceed to the second intervention if (1) their dyspnea level was >/= baseline dyspnea level-1, or (2) their dyspnea level was >/= 3/10 after one hour.
Time Frame: Minimally 1 hour, up to 5 hours
Measure: Number; unit: Participants
Arm/Group | Group 1: BiPAP Then Vapotherm | Group 2: Vapotherm Then BiPAP
Number analyzed (Participants) | 10 | 13
Participants
  Completed washout period | 7 | 10
  Completed second intervention | 3 | 5

2. Primary Outcome: Effects of BIPAP and VapoTherm Device on Severity of Dyspnea as Measured by the Numeric Rating Scale
Description: Dyspnea, a subjective sensation experienced by participants, was assessed with the numeric rating scale (NRS) before and after each 2 hour intervention. The NRS is a validated 11-point scale ranging from 0 (no dyspnea) to 10 (worst dyspnea). Participants received either (1) 2 hours of HFO followed by a variable washout period and then 2 hours of BiPAP or (2) 2 hours of BiPAP followed by a variable wash-out period and then 2 hours of HFO.
Time Frame: Up to 5 hours, baseline/enrollment to 5 hours (2 hours for each treatment with variable wash-out period)
Population: One participant assigned to receive BiPAP was mistakenly started on Vapotherm (High Flow Oxygen = HFO), and was reported here in the HFO group.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1: BiPAP Then Vapotherm | Group 2: Vapotherm Then BiPAP
Number analyzed (Participants) | 14 | 16
units on a scale
  Dyspnea NRS at the time of enrollment | 7 [5 to 8] | 6 [4 to 8]
  Dyspnea NRS after intervention | 3.4 [1.8 to 5.0] | 4.2 [3.1 to 5.4]

ADVERSE EVENTS:
Time Frame: Study participation time was approximately 5 hours, from enrollment till second air delivery treatment completed. Total study period was 2 years and 4 months.
Description: Adverse events were recorded at enrollment before measurements/interventions were completed while participants were on baseline oxygen. No adverse events were reported/associated with device use during treatment periods therefore reporting was provided by group assignment rather than treatment received.
Groups:
- Group1: BiPAP Then Vapotherm: Bilevel positive airway pressure device (BiPAP) air delivery then Vapotherm device air delivery.
- Group 2: Vapotherm Then BiPAP: Vapotherm device air delivery then Bilevel positive airway pressure device (BiPAP) air delivery.
Arm/Group | Group1: BiPAP Then Vapotherm | Group 2: Vapotherm Then BiPAP
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group1: BiPAP Then Vapotherm (N=15) | Group 2: Vapotherm Then BiPAP (N=15)
Dry eyes before intervention (Eye disorders) | 1 (1) | 3 (3)
Eye irritation before intervention (Eye disorders) | 1 (1) | 3 (3)
Anxiety before intervention (Psychiatric disorders) | 2 (2) | 1 (1)
Moist nose before intervention (General disorders) | 2 (2) | 2 (2)
Prong Uncomfortable before intervention (General disorders) | 2 (2) | 2 (2)
Stomach bloating before intervention (Gastrointestinal disorders) | 1 (1) | 3 (3)
Suffocating before intervention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Trouble drinking before intervention (Gastrointestinal disorders) | 1 (1) | 0 (0)
Trouble eating before intervention (Gastrointestinal disorders) | 2 (2) | 5 (5)
Trouble sleeping before intervention (General disorders) | 2 (2) | 7 (7)
Trouble talking before intervention (Social circumstances) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No